CLINICAL TRIAL: NCT04569240
Title: Accuracy of the Dexcom G6 Continuous Glucose Monitoring System Following Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Principal Investigator, M. Cecilia Lansang, MD, Staff Physician, Director - Endocrinology Main Campus, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-698
Record Dates: First submitted 2020-09-08; First posted 2020-09-29 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Surgery--Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Dexcom G6 continuous glucose monitor (Other): All patients will have a Dexcom G6 continuous glucose monitor placed pre-operatively. The glucose readings will be collected for 10 days or upon discharge from the ICU and data will be compared with arterial blood glucose readings or venous Accu-Check Inform II glucose readings
  Interventions: Device: Dexcom G6 continuous glucose monitor

INTERVENTIONS:
Device: Dexcom G6 continuous glucose monitor — Dexcom G6 continuous glucose monitor will be applied to the upper outer arm before cardiovascular surgery. Data will be collected for 10 days or upon discharge from the ICU.

SUMMARY:
This is a prospective longitudinal study to study the agreement between a novel continuous glucose monitoring system (CGMS) versus current blood glucose monitoring.

Subjects in this study will have their blood glucose measured regularly every 1-3 hours with current methods in the cardiovascular intensive care unit (CVICU), and by point of care glucose using the Accuchek Inform II on the regular floors, and the CGMS at the same time will be captured. Subjects will have measurements taken throughout their stay in the CVICU and on the regular floors.

DETAILED DESCRIPTION:
Maintaining tight blood glucose control following surgery is imperative to reducing infections and neurologic dysfunction. This requires frequent blood sampling while in the intensive care unit, leading to increased waste of blood and utilizing time and resources to collect samples and wait for results. Additionally, when on the regular floors, frequent point of care fingersticks for glucose levels are needed for therapeutic intervention.

Continuous glucose monitoring systems (CGMS) are now available for ambulatory use in patients with diabetes. The potential of using such a system in the hospital, including during the postoperative critical care setting and upon transfer to the regular floor, may reduce personnel burden, produce rapid results, and decrease blood waste. However, these systems have not yet been validated for hospital use.

This is a prospective longitudinal study to study the agreement between a novel continuous glucose monitoring system (CGMS) versus current blood glucose monitoring.

Subjects in this study will have their blood glucose measured regularly every 1-3 hours with current methods in the CVICU, and by point of care glucose using the Accuchek Inform II on the regular floors, and the CGMS at the same time will be captured. Subjects will have measurements taken throughout their stay in the CVICU and on the regular floors. Agreement and correlation between systems will be calculated, and error will be classified using the Surveillance Error grid. The proportion of errors of at least moderate risk will be calculated.

Subject characteristics including demographics, comorbidities and baseline disease severity will be summarized using means and standard deviations for continuous measures and frequencies and percentages for categorical factors. To evaluate agreement between methods, concordance correlation coefficients will be calculated, using the method that adjusts for repeated measures as described by King and implemented in software by Carrasco. Analysis will be performed overall, and then stratifying by type of current measure, if the type of measurement varies across settings. Correlations will be calculated using the methods described by Bland and Altman and implemented by Bakdash and Marusich. Differences will also be evaluated for errors according to the Surveillance Error Grid. Rates of moderate or more severe errors will be calculated. For each measure above, 95% confidence intervals will be calculated, accounting for the clustering within subject.. Analyses will be performed using SAS software (version 9.4; Cary, NC) and R software (version 3.5; Vienna Austria).

Glucose readings obtained from the CGMS will be compared with

1. blood glucose from the arterial blood gas (ABG) or peripheral/central venous catheter if arterial catheter not in use (standard of care in CVICU) while patients are in the CVICU
2. fingerstick point of care (POC) glucose when patients are on the regular floors

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and above
* Planned cardiovascular surgery
* Planned admission to Cleveland Clinic Main Campus J5 or J6 or Q5 cardiovascular ICU (CVICU) post-operatively
* With or without known diabetes; if with known diagnosis of diabetes, diabetes can be type 1, type 2, or secondary

Exclusion Criteria:

* Allergy to the material of the CGMS or the adhesive to be used
* Skin conditions precluding the use of the CGMS
* Pregnancy
* Other conditions that investigators deem inappropriate for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-01-20 (Actual); Study Completion 2024-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. Cecilia Lansang, MD, MPH, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] King TS, Chinchilli VM, Carrasco JL. A repeated measures concordance correlation coefficient. Stat Med. 2007 Jul 20;26(16):3095-113. doi: 10.1002/sim.2778. PMID 17216594
- [Background] Carrasco JL, Phillips BR, Puig-Martinez J, King TS, Chinchilli VM. Estimation of the concordance correlation coefficient for repeated measures using SAS and R. Comput Methods Programs Biomed. 2013 Mar;109(3):293-304. doi: 10.1016/j.cmpb.2012.09.002. Epub 2012 Sep 29. PMID 23031487
- [Background] Bland JM, Altman DG. Calculating correlation coefficients with repeated observations: Part 1--Correlation within subjects. BMJ. 1995 Feb 18;310(6977):446. doi: 10.1136/bmj.310.6977.446. No abstract available. PMID 7873953
- [Background] Bakdash JZ, Marusich LR. Repeated Measures Correlation. Front Psychol. 2017 Apr 7;8:456. doi: 10.3389/fpsyg.2017.00456. eCollection 2017. PMID 28439244
- [Background] Klonoff DC, Lias C, Vigersky R, Clarke W, Parkes JL, Sacks DB, Kirkman MS, Kovatchev B; Error Grid Panel. The surveillance error grid. J Diabetes Sci Technol. 2014 Jul;8(4):658-72. doi: 10.1177/1932296814539589. Epub 2014 Jun 13. PMID 25562886

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dexcom G6 continuous glucose monitor
Started | 40
Completed | 29
Not Completed | 11

BASELINE CHARACTERISTICS:
Arm/Group | Dexcom G6 Continuous Glucose Monitor
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data was not collected for all participants
  Participants
    number analyzed (Participants) | 24
    Female | 7
    Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Data was not collected on 4 participants
  Participants
    number analyzed (Participants) | 25
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 1
    White | 23
    More than one race | 0
    Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] — Population: Data was not collected for all participants
  kg/m2
    number analyzed (Participants) | 25
    (all) | 30.2 (4.9)
Participants with diabetes [Count of Participants; unit: Participants] — Diabetes diagnosis can be type 1, type 2, or secondary (such as due to glucocorticoids or pancreatitis) Population: Data was not collected for all participants
  Participants
    number analyzed (Participants) | 25
    (all) | 25
Surgery [Count of Participants; unit: Participants] — Population: Data was not collected for all participants
  Participants
    number analyzed (Participants) | 25
    aortic valve replacement/ascending | 9
    Bentall | 2
    coronary artery bypass graft | 4
    coronary artery bypass graft/extended | 6
    mitral valve replacement | 1
    Myectomy | 1
    Pericardiectomy | 1
    right ventricular assist device | 1
Intravenous insulin use during surgery [Count of Participants; unit: Participants] — Population: Data was not collected for all participants
  Participants
    number analyzed (Participants) | 25
    (all) | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Matching Glucose Measurements (CGM Versus Blood Glucose Measurements)
Description: Glucose readings from the Dexcom continuous glucose monitor compared with blood glucose from the arterial blood gas (ABG) or peripheral/central venous catheter
Time Frame: Up to 10 days
Population: Total matched observations vs. matched glucose measures
Measure: Number; unit: matched clinical glucose measure
Units Other Than Participants: Total matched observations
Arm/Group | Dexcom G6 continuous glucose monitor
Number analyzed (Participants) | 29
Number analyzed (Total matched observations) | 817
matched clinical glucose measure | 817

2. Primary Outcome: Glucose Readings From Continuous Glucose Monitor (CGM) Versus Point of Care Glucose
Description: Glucose readings in mg/dL from the Dexcom continuous glucose monitor (CGM) will be compared with fingerstick point of care glucose levels in mg/dL
Time Frame: up to 10 days
Population: matched clinical glucose measure
Measure: Number; unit: matched clinical glucose measure
Units Other Than Participants: Total matched glucose measures
Arm/Group | Dexcom G6 continuous glucose monitor
Number analyzed (Participants) | 29
Number analyzed (Total matched glucose measures) | 817
matched clinical glucose measure
  Total matched observations | 817
  Matched fingerstick measures | 280

3. Other Pre Specified Outcome: Blood Volume Waste by Arterial Blood Gas
Description: Blood sample amounts in milliliters required for measurement of glucose by arterial blood gas
Time Frame: Up to 10 days
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Blood Volume Waste by Fingerstick
Description: Blood sample amounts in milliliters required for measurement of glucose by fingerstick
Time Frame: Up to 10 days
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Cost Savings:
Description: Cost of CGMS device including sensor, transmitter versus cost of doing an ABG to obtain glucose levels (CVICU stay), and versus the cost of Accu-chek Inform II meter, test strips, and lancets
Time Frame: Up to 10 days
Population: No Cost saving analysis was performed
Arm/Group | Dexcom G6 continuous glucose monitor
Number analyzed (Participants) | 0

6. Other Pre Specified Outcome: Time Savings
Description: time it takes to perform and time it takes to have results based on an ABG or fingerstick POC on Accu-check Inform II
Time Frame: Up to 10 days
Population: This outcome measure was not analyzed
Arm/Group | Dexcom G6 continuous glucose monitor
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Dexcom G6 continuous glucose monitor
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 3/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dexcom G6 continuous glucose monitor (N=29)
Dexcom site pain (Musculoskeletal and connective tissue disorders) | 3 — Numbness and pain on the same arm the device was placed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-12): https://cdn.clinicaltrials.gov/large-docs/40/NCT04569240/Prot_SAP_000.pdf